CLINICAL TRIAL: NCT03639428
Title: Pharmacokinetic Evaluation of MDZ028 After Single Administration of a New Oral Form, at the Time of Anesthetic Premedication in Children.
Brief Title: Pharmacokinetic Evaluation of MDZ028
Acronym: MIDAZOLAM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI10-PR-DUPONT
Record Dates: First submitted 2018-08-01; First posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Midazolam
Keywords: pharmacokinetics; child; cyclodextrin; moderate sedation
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 6 - 23 months: 8 infants between 6 and 23 months received a single 0.3mg/kg midazolam dose of ADV6209
  Interventions: Drug: Midazolam
- 2-11 years: 17 children between 2 and 11 years received a single 0.3mg/kg midazolam dose of ADV6209
  Interventions: Drug: Midazolam
- 12-17 years: 12 adolescents between 12 and 17 years received a single 0.3mg/kg midazolam dose of ADV6209
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Midazolam — All subjects received a sigle 0.3mg/kg midazolam dose os ADV6209
  Other Names: midazolam dose of ADV6209

SUMMARY:
Plasma concentration data were collected from 37 paedriatic patients and 12 healthy adults recruited in a single dose, open-label phase II pharmacokinetic study and in a single dose, randomised, open-label two-peiod crossover bioavailability study, respectively. Data were analysed using non-linear mixed effect modeling.

DETAILED DESCRIPTION:
In the absence of a licensed formulation in many countries worldwide, ADV6209, an innovative 2mg/ml oral solution of midazolam containing cyclodextrin, has been developed for moderate sedation in paediatric patients. Population pharmacokinetics for ADV6209 is reported.

Plasma concentration data were collected from 37 paedriatic patients and 12 healthy adults recruited in a single dose, open-label phase II pharmacokinetic study and in a single dose, randomised, open-label two-peiod crossover bioavailability study, respectively. Data were analysed using non-linear mixed effect modeling. Plasma concentrations of midazolam were discribed by a two-compartement model. An additional one-compartement model was added for a α-hydroxymidazolam.

ELIGIBILITY:
Inclusion Criteria:

* Child (boy or girl) for whom surgery under general anesthesia is scheduled.
* Child aged 6 months to 17 years old.
* Child with a body mass index between the 3rd and 97th percentile.
* Child with ASA (American Society of Anesthesiology) status of I or II. Young girl of childbearing age (ie after puberty) and sexually active to have a result negative to the pregnancy test.
* Child whose parents / legal representative (s) agree to sign a consent form.
* Child whose opinion / agreement was / tried to be collected.
* Child and parents / legal representative (s) being ready and able to participate in the study, understanding and undertaking to respect the study procedures throughout the duration of the study.
* Child enrolled in a social security scheme.

Exclusion Criteria:

* Child with midazolam allergy, benzodiazepine hypersensitivity or hypersensitivity known to one of the excipients of the formulation of the study.
* Child with respiratory disease (severe respiratory failure, acute respiratory depression).
* Child with heart disease.
* Child with gastrointestinal disorders that may affect absorption or gastroesophageal reflux.
* Child with growth disorders or abnormal weight-of-weight.
* Child taking Cytochrome P450 Interactions Within 60 Days of Inclusion in the study.
* Child with kidney failure, liver failure, history of myasthenia gravis, or neurological disease.
* Pregnant or lactating girl.
* Child who has a known human immunodeficiency virus (HIV) infection, or active hepatitis B, or active hepatitis C.
* A child who could present any condition that may prevent his participation in the study, according to the judgment of the investigator.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The planned enrollment is 36 children, stratified in two groups: 24 children between 6 months and 11 years, and 12 children between 12 and 17 years. Age is considered in years past by the date of inclusion. Children aged between 6 months and 11 years old should be homogenous in both age groups 6-23 months and 2-11 years. For example, at least 4 children in the 6-23 month age group will be recruited.
  Children likely to be included will be hospitalized in the pediatric surgery department at Amiens University Hospital.
  Children who will be included in this study will not be able to participate in another study within 3 months of their inclusion in this study.
Sampling Method: Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2011-06-23 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic analysis of the oral solution of midazolam (ADV6209) | 1 day
  The Aim of the study was to assess the pharmacokinetic analysis of an oral solution of midazolam (ADV6209) oral formulation in paedriatic patients from 6 months to 18 years ols in order to support dosing recommendations. All subjects received a single 0.3mg/kg midazolam dose of ADV6209, without exceeding a total dose of 10 mg.Population pharmacokinetic modelling was performed to characterise the concentration-time course of midazolam and its main active metabolite, and to evaluate the changes in clearance and volume of distibution in the different age groups.

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Dupont, MD, PhD, Principal Investigator — CHU AMIENS

IPD SHARING:
Plan to Share IPD: No